CLINICAL TRIAL: NCT03900767
Title: Multi-Level Interventions for Increasing Tobacco Cessation at Federally Qualified Health Clinics (FQHCs)
Brief Title: Strategies to Connect Patients at Federally Qualified Health Clinics With Evidence Based Tobacco Cessation Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Utah (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, David Wetter, Principal Investigator, University of Utah
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HCI111985; NCI-2019-00502 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HCI111985 (Other: Huntsman Cancer Institute/University of Utah)
Record Dates: First submitted 2019-03-11; First posted 2019-04-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Current Smoker; Tobacco Smoking; Tobacco Use
Keywords: Text Messaging; Underserved Population; Underserved; Utah; Tobacco Cessation
MeSH Terms: conditions — Tobacco Smoking; Tobacco Use; Tobacco Use Cessation | interventions — Smoking Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Clinic-Level (Experimental): Clinics will receive the AAC intervention consisting of an EHR-based point of care alert that prompts clinic staff to Ask every patient about tobacco use, Advise tobacco using patients to quit, and Connect interested tobacco users to the Utah Tobacco Quit Line
  Assigned Interventions = Electronic Health Record intervention AAC
  Interventions: Other: Electronic Health Record intervention
- Phase I Group I (Continued EHR and text messages) (Experimental): Patients receive a weekly text message for one month followed by a monthly text message over the next 5 months (i.e., 6 months of text messages following each tobacco users' clinic visit). All messages will include a motivational message, the Quit Line website, the Quit Line phone number, and simple two-touch response that directly connects interested tobacco users to the Quit Line.
  Interventions: Other: Electronic Health Record intervention; Behavioral: Smoking Cessation Intervention; Behavioral: Telephone-Based Intervention
- Phase I Group II (Continued clinic-level EHR intervention only) (Experimental): Patients receive continued clinic level EHR intervention only (CO).
  Interventions: Other: Electronic Health Record intervention; Behavioral: Smoking Cessation Intervention
- Phase II Group I (Text messages, Counseling call) (Experimental): Patients receive a monthly text message plus 2 brief telephone calls from patient navigators/health educators for 6-12 months following each tobacco user's clinic visit.
  Interventions: Other: Electronic Health Record intervention; Behavioral: Smoking Cessation Intervention; Behavioral: Telephone-Based Intervention
- Phase II Group II (Text messages continued) (Experimental): Patients receive a monthly text message for 6-12 months following each tobacco user's clinic visit that includes a simple one-touch response to directly connect to the Quitline.
  Interventions: Other: Electronic Health Record intervention; Behavioral: Smoking Cessation Intervention; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Electronic Health Record intervention — AAC
Behavioral: Smoking Cessation Intervention — Receive standard Utah Quitline treatment
  Other Names: Smoking and Tobacco Use Cessation Interventions
  Arms: Phase I Group I (Continued EHR and text messages); Phase I Group II (Continued clinic-level EHR intervention only); Phase II Group I (Text messages, Counseling call); Phase II Group II (Text messages continued)
Behavioral: Telephone-Based Intervention — Receive text messages
  Arms: Phase I Group I (Continued EHR and text messages); Phase II Group I (Text messages, Counseling call); Phase II Group II (Text messages continued)
Behavioral: Telephone-Based Intervention — Receive phone calls
  Arms: Phase II Group I (Text messages, Counseling call)

SUMMARY:
This trial aims to connect tobacco using patients of Community Health Centers (CHCs) and Federally Qualified Health Centers (FQHCs) with evidence-based treatment to help them quit. The trial will evaluate multiple strategies, that target both clinics and for patients, to increase the number of patients who enroll in Utah Tobacco Quit Line treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate clinic and patient level interventions with respect to increasing the reach of evidence-based treatment for tobacco use (delivered via the Utah Quitline).

II. To evaluate clinic and patient level interventions with respect to increasing the impact of Quitline treatment. Impact is defined as Reach X Efficacy. In calculating impact, efficacy is defined as the proportion of smokers who enroll in Quitline delivered treatment that successfully quit.

III. To evaluate characteristics of both clinics and patients that may influence tobacco use outcomes.

OUTLINE:

CLINIC-LEVEL INTERVENTION

All clinics will receive a clinic-level intervention of Ask Advise Connect (AAC). AAC consists of an electronic health record (EHR) intervention that utilizes the EHR to facilitate clinic staff to Ask patients about tobacco use, Advise patients to quit using tobacco, and directly and electronically Connect patients to the Utah Tobacco Quit Line.

PHASE I (PATIENT-LEVEL): Patients who do not enroll in the Quit Line following the clinic visit will be eligible for Phase 1 randomization to receive either TM or continue with the EHR Condition Only (CO).

GROUP I: Patients receive a Text Message (TM) weekly for one month followed by a monthly text message with a one-touch response to connect to the Quit Line over the next 5 months (i.e., 6 months of text messages following the clinic visit).

GROUP II: Patients receive continued clinic level EHR intervention only (CO).

PHASE II (Patient-level): Nonresponders (i.e., did not enroll in Quit Line treatment at 6 months) in Group 1 of Phase I (TM/CO) will be randomized to 1 of 2 groups:

GROUP I: Patients will continue to receive text messages (motivational messaging with simple touch response to connect directly to the Quit Line) plus 2 brief telephone calls from health coaches for 6-12 months following the clinic visit. Brief telephone coaching calls will be conducted using Motivation and Problem Solving (MAPS) for a TM+MAPS condition.

GROUP II: Patients continue to receive a monthly text message with a one-touch response to directly connect to the Quit Line during months 6-12 following the clinic visit, i.e., text message continued (TM-Cont).

Roughly twelve months after the clinic visit, eligible patients will be invited to complete a 12-month survey on quality of life and abstinence assessments.

A saliva kit will be sent to 300 randomly selected patients who indicate abstinence at the 12-month follow-up and agree to the saliva sample.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be current tobacco users.
* Participants who speak English or Spanish.
* Participants will have a working cellphone that can accept texts and calls.
* Participants who present at participating community health center (CHC) clinics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12009 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Reach | Up to 12 months
  Defined as the proportion of tobacco users who enter Quitline treatment.
Impact | At 12 months
  Defined as reach x efficacy. Efficacy is defined as the proportion of tobacco users entering Quitline treatment who quit (i.e., achieve abstinence).
Abstinence from tobacco use | At 12 months
  Abstinence assessments are based on recommendations for cessation induction trials (i.e., 7 and 30 day point prevalence abstinence).
Health-related quality of life | At 12 months
  Assessed with the Short Form Health Survey (SF-12)

SECONDARY OUTCOMES:
Abstinence from tobacco use (biochemical validation) | At 12 months
  We will randomly select a subset of participants who report abstinence at 12 months follow-up survey to complete biochemical validation of abstinence via saliva samples. The saliva sample will be used to test for cotinine, a metabolite of nicotine.

CONTACTS AND LOCATIONS:
Overall Officials: David Wetter, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez ME, Schlechter CR, Del Fiol G, Gibson B, Kawamoto K, Siaperas T, Pruhs A, Greene T, Nahum-Shani I, Schulthies S, Nelson M, Bohner C, Kramer H, Borbolla D, Austin S, Weir C, Walker TW, Lam CY, Wetter DW. QuitSMART Utah: an implementation study protocol for a cluster-randomized, multi-level Sequential Multiple Assignment Randomized Trial to increase Reach and Impact of tobacco cessation treatment in Community Health Centers. Implement Sci. 2020 Jan 30;15(1):9. doi: 10.1186/s13012-020-0967-2. PMID 32000812

DOCUMENTS (1):
  • Informed Consent Form (2022-09-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT03900767/ICF_000.pdf